CLINICAL TRIAL: NCT01327599
Title: Assessing the Efficacy and Tolerability of Changing to DUOTRAV® (Travoprost 0.004%/Timolol 0.5% BAK-Free Fixed Combination), as Replacement Therapy in Patients Previously on Bimatoprost 0.03%/Timolol 0.5% Therapy (Fixed or Unfixed)
Brief Title: Efficacy of Changing to DUOTRAV® From Prior Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-10-272; 2011-000161-13 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension; Pigment Dispersion Glaucoma
Keywords: Open-angle glaucoma; Ocular hypertension; Pigment dispersion glaucoma; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Timolol; Ophthalmic Solutions; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DUOTRAV® (Experimental): Travoprost 0.004%+Timolol 0.5% ophthalmic solution, 1 drop to the study eye(s) once a day at 8:00 PM for 12 weeks
  Interventions: Drug: Travoprost 0.004%+Timolol 0.5% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004%+Timolol 0.5% ophthalmic solution — Fixed dose combination topical ocular agent preserved with polyquaternium-1 (POLYQUAD)
  Other Names: DUOTRAV®

SUMMARY:
The purpose of this study was to assess the efficacy and tolerability of changing to DUOTRAV® from prior bimatoprost 0.03%/timolol 0.5% pharmacotherapy in subjects with open-angle glaucoma or ocular hypertension having uncontrolled intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, open-angle or pigment dispersion glaucoma in at least one eye.
* Stable IOP-lowering regimen of bimatoprost 0.03%/timolol 0.5% therapy (either administered concomitantly or in a fixed combination) within 4 weeks prior to the screening visit.
* IOP considered to be safe (in the opinion of the investigator), in both eyes, to assure clinical stability of vision and the optic nerve throughout the study period.
* IOP between 19 to 35 mmHg (at any time of the day) in at least one eye (which would be designated as the study eye).
* Willing to discontinue the use of all other ocular hypotensive medication(s) prior to receiving the study medication for the entire course of the study.
* Able to follow instructions and willing and able to attend all study visits.
* Best corrected visual acuity of 6/60 (20/200 Snellen, 1.0 LogMAR) or better in each eye.
* Sign informed consent.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any component of DuoTrav® that is deemed clinically significant in the opinion of the Principal Investigator.
* Corneal dystrophies in either eye.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Bronchial asthma or a history of bronchial asthma, bronchial hyper reactivity, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* History of severe allergic rhinitis.
* A condition, which in the opinion of the Principal Investigator, would interfere with optimal participation in the study, or which would present a special risk to the subject.
* Participation in any other investigational study within 30 days prior to the Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Durier, Pharm.D, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 study centers in France and 3 study centers in Germany.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | DUOTRAV®
Started | 60
Completed | 57
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Could Not Attend Visit | 1
Not completed — Withdrawal of Consent | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all participants who received study medication and had at least one on-therapy study visit (Intent-to-treat).
Arm/Group | DUOTRAV®
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in IOP at Week 12 in Subjects Using Ganfort® at Baseline
Description: IOP (fluid pressure in the eye) was measured with Goldmann applanation tonometry. A positive number change from baseline indicates an increase in intraocular pressure, which may be a risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye was chosen as the study eye, and only the study eye was used for analysis.
Time Frame: Week 12
Population: All subjects using Ganfort at baseline who received study medication and attended Week 12 visit.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | DUOTRAV®
Number analyzed (Participants) | 55
millimeters mercury (mmHg)
  Baseline (Day 1) | 20.0 (1.0)
  Change from baseline at Week 12 | -3.8 (1.9)

2. Secondary Outcome: Mean Change From Baseline in Ocular Surface Disease Index (OSDI) Score at Week 12 in Subjects Using Ganfort® at Baseline
Description: The OSDI is a 12-item quality of life questionnaire designed to assess ocular surface symptoms, their severity, and their impact on the subject's ability to function. Each item was scored by the subject on a 0-4 Likert-type scale (0=None, 4=All of the Time), with a resultant overall score of 0-100 (0=no disability, 100=complete disability). A negative number change from baseline represents a perceived improvement in ocular health.
Time Frame: Week 12
Population: ITT: All subjects using Ganfort at baseline who received study medication and had at least one on-therapy study visit, minus missing responses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DUOTRAV®
Number analyzed (Participants) | 57
Units on a scale
  Baseline (Day 1) | 14.9 (10.9)
  Change from Baseline at Week 12 | -3.6 (6.5)

3. Secondary Outcome: Mean Change From Baseline in Ocular Hyperemia Score at Week 12 in Subjects Using Ganfort® at Baseline
Description: Ocular hyperemia (visible eye redness) was assessed during slit lamp examination and graded on a 5-point scale (0=none, 4=severe). A positive number change from baseline indicates an increase in ocular redness. One eye was chosen as the study eye, and only the study eye was used for analysis.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DUOTRAV®
Number analyzed (Participants) | 57
units on a scale | -0.1 (0.7)

4. Secondary Outcome: Percentage of Subjects Who Reach Target IOP of ≤ 18 mmHg in Subjects Using Ganfort® at Baseline
Description: IOP (fluid pressure in the eye) was measured with Goldmann applanation tonometry. An increase in intraocular pressure may be a risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye was chosen as the study eye, and only the study eye was used for analysis.
Time Frame: Week 4, Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | DUOTRAV®
Number analyzed (Participants) | 57
percentage of participants
  Week 4 | 78.6
  Week 12 | 85.5

5. Secondary Outcome: Mean Change From Baseline in IOP at Week 4 in Subjects Using Ganfort® at Baseline
Description: as for outcome 1
Time Frame: Week 4
Population: All subjects using Ganfort at baseline who received study medication and attended Week 4 visit.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | DUOTRAV®
Number analyzed (Participants) | 57
millimeters mercury (mmHg)
  Baseline (Day 1) | 20.1 (1.1)
  Change from Baseline at Week 4 | -3.8 (2.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (1 year, 3 months). An adverse event was defined as any untoward medical occurrence in a subject administered a study treatment regardless of causal relationship.
Description: Adverse events were collected spontaneously from the subjects and systematically by inquiry and review of protocol-specific ocular or systemic parameters evaluated during the study. This reporting group includes all participants who received study medication.
Arm/Group | DUOTRAV®
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
France: All results obtained during this study are the property of the Sponsor. All information given to the investigators must remain confidential and cannot be used outside the framework of this study. Germany: Investigators can publish results 12 months after the Sponsor's final evaluation of the data. The Sponsor is entitled to request a delay of such publication due to business or operational reasons.